CLINICAL TRIAL: NCT06678568
Title: The Optimized Follow-up Protocol for Pediatric Metaphyseal Forearm Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nonticha Thanthong (Other)
Responsible Party: Sponsor-Investigator, Nonticha Thanthong, Sponsor Investigator, Ramathibodi Hospital
Organization: Ramathibodi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MURA2024/689
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Wrist Fracture
Keywords: metaphyseal forearm fracture; loss of reduction; follow-up protocol; wrist fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The standard follow-up protocol (No Intervention): follow-up and film every week at hospital
- The optimized follow-up protocol (Experimental): follow-up and film every week at hospital except the 3rd week is telemedicine follow-up
  Interventions: Other: telemedicine follow-up in 3rd week

INTERVENTIONS:
Other: telemedicine follow-up in 3rd week — Intervention group will be appointed with telemedicine follow-up in 3rd week after injury, instead of hospital follow-up visit.
  Arms: The optimized follow-up protocol

SUMMARY:
The randomized controlled study which compare radiologic outcomes (loss of reduction rate) and complications in pediatric patients with displaced metaphyseal forearm fractures who underwent conservative treatment. The patients were assigned in two different follow-up protocols. In the control group, the patients will go to hospital for follow-up visit and film every week until 4th week after injury. In the intervention group, the patients will go to hospital for follow-up visit every week except in the 3rd week after injury they will be gotten telemedicine follow-up.

DETAILED DESCRIPTION:
Randomization of patients for 2 different follow-up protocols

Objective: to compare loss of reduction rate by angulation measurement and prevalence of complications in patients with displaced metaphyseal forearm fractures who underwent conservative treatment.

Method:

Patients will be randomly assigned to one of two groups using various block computerized randomization. Randomization will be performed using STATA version 16.0, Statacorp, College Station, Texas, USA

Interventions:

Group 1 (control group): The patients will go to hospital for follow-up visit and film every week until 4th week after injury.

Group 2 (intervention group): The patients will go to hospital for follow-up visit every week except in the 3rd week after injury they will be gotten telemedicine follow-up.

Treatment Allocation and concealment:

A randomization will prepare with sealed envelopes containing assigned follow-up protocols for each patient.

The envelopes will be labeled with the study ID.

Blinding:

Because of the two different of follow-up protocol, we cannot blind the protocol from participants, physicians and assessors.

Outcomes:

1. Primary outcome is loss of reduction rate using angulation measurement. The definition of loss of reduction angulation is angulation which is more than 10 degree in coronal view or more than 20 degree in sagittal view. Angulation measurement will be measured in bisector between longitudinal axis and center of diaphysis. Angulation will be measured by two physicians and two times using PACS (Picture Archiving and Communication System) in Ramathibodi hospital.
2. Secondary outcomes are other complications such as malunion, nonunion, joint stiffness and cast problem

Statistical Analysis Plan:

Data will be recorded in Microsoft Excel and imported to STATA version 16.0 for re-check.

For continuous data, use mean and standard deviation (S.D.) For categorical data, use frequency and percentage For comparing non-normal distribution between group, use Mann-Whitney test and for continuous data, use Fisher's exact test Define the Statistical significant is p-value < 0.05 Data analysis will be performed with STATA version 16.0, Statacorp, College Station, Texas, USA.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-12 years
* Patients with distal metaphyseal forearm fractures in Ramathibodi hospital and Chakri Naruebodindra Medical Institute
* Presented to hospital within 72 hours of injury

Exclusion Criteria:

* Open fracture
* Operative treatment at 1st visit
* Neurovascular injury
* Polytraumatized patient
* Ipsilateral fracture of upper limb
* History of previous surgery in the affected arm
* Metabolic bone disease

Max Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-11-05 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
loss of reduction rate | From enrollment to the end of treatment at 4 weeks
  Angulation is more than 10 degree in coronal view or more than 20 degree in sagittal view

SECONDARY OUTCOMES:
Complications | From enrollment to the end of treatment at 4 weeks
  Number of Participants with malunion, nonunion, joint stiffness and cast problem

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No